CLINICAL TRIAL: NCT00783965
Title: A Phase II Randomized, Double-Blind, Vehicle-Controlled, Crossover Clinical Trial of Tazarotene 0.1% and Vehicle Cream Each Applied Once-Daily for 12 or 24 Months in Subjects With Basal Cell Nevus Syndrome
Brief Title: Topical Tazarotene in Treating Patients With Basal Cell Skin Cancer and Basal Cell Nevus Syndrome on the Chest and Back
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR0000618240; 5R01CA109584-05 (NIH); U19CA081888 (NIH)
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-01

CONDITIONS: Skin Carcinoma
Keywords: nevoid basal cell carcinoma syndrome; basal cell carcinoma of the skin
MeSH Terms: conditions — Basal Cell Nevus Syndrome; Carcinoma, Basal Cell | interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients apply 0.1% tazarotene cream on months 0-12 and vehicle (placebo) on months 13-36 once daily to the chest.
  Interventions: Drug: tazarotene; Other: placebo
- Arm II (Experimental): Patients apply, vehicle (placebo) on months 0-12 and 0.1% tazarotene cream on months 13-36 once daily to the chest.
  Interventions: Drug: tazarotene; Other: placebo

INTERVENTIONS:
Drug: tazarotene — Applied to the skin
  Other Names: tazorac
Other: placebo — Applied to the skin
  Other Names: vehicle

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as tazarotene, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This randomized phase II trial is comparing two different schedules of topical tazarotene and topical placebo to see how well they work in treating patients with basal cell skin cancer and basal cell nevus syndrome on the chest.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To expand and refine chemopreventive strategies in individuals with basal cell nevus syndrome (BCNS) on the chest and back, who are at high risk for the development of basal cell carcinomas (BCCs).
* To determine whether tazarotene 0.1% cream applied to the chest for two years will reduce the numbers of basal cell carcinomas (BCCs) observed, as compared to the number expected, based on changes in BCC numbers observed during months 0-12.

Secondary

* To compare the difference in total BCC burden (measured as the total lesion surface area) between chest and back over various time points and aggregated intervals of interest.
* To determine whether there are any detectable wash-in or wash-out periods for the tazarotene effects.
* Explore the use of a random effects model for longitudinal analysis of total lesions over time.

OUTLINE: This is a multicenter study. Patients are randomized into 1 of 2 arms.

* Arm I: Patients apply 0.1% tazarotene cream on months 0-12 and vehicle (placebo) on months 13-36 once daily to the chest in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients apply vehicle (placebo) on months 0-12 and 0.1% tazarotene cream on months 13-36 once daily to the chest in the absence of disease progression or unacceptable toxicity.

Treated chest and untreated back is evaluated at 3 month intervals for 36 months.

ELIGIBILITY:
List of Inclusion Criteria:

1. Study subjects must have at least one basal cell carcinoma ≥ 3mm in diameter (target lesion) on any area of the skin except the face, chest, and back (and not impinging on vital sites) diagnosed clinically by a Study Investigator at the baseline visit.
2. Study subjects must meet diagnostic criteria for basal cell nevus syndrome including major criterion #1 plus one additional major criterion or two of the minor criteria outlined in Table I. A first degree relative would satisfy BCNS diagnostic criteria with any two major criteria or any single major plus two minor criteria.

Table I. BCNS Diagnostic Criteria

Major criteria

1. More than 2 BCCs or one under the age of 20 years
2. Odontogenic keratocysts of the jaw proven by histology
3. Three or more palmar and/or plantar pits
4. Bilamellar calcification of the falx cerebri (if less than 20 years old)
5. Fused, bifid, or markedly splayed ribs.
6. First degree relative with basal cell nevus syndrome (BCNS)
7. PTCH1 gene mutation in normal tissue*

Minor criteria

1. Macrocephaly determined after adjustment for height
2. Congenital malformations: cleft lip or palate, frontal bossing, "coarse face."
3. Skeletal abnormalities: Sprengel deformity, marked pectus deformity
4. Radiological abnormalities: bridging of the sella turcica, vertebral anomalies such as hemivertebrae, fusion or elongation of the vertebral bodies.
5. Ovarian fibroma
6. Medulloblastoma

3.The subject is from 18-75 years of age, inclusive.

4. If the subject is female and of child-bearing potential (women are considered not of childbearing potential if they are at least 2 years post-menopausal and/or surgically sterile), she:

i. has been using adequate contraception (abstinence, IUD, birth control pills, or spermicidal gel with diaphragm or condom) since her last menses and will use adequate contraception during the study, and ii. is not lactating, and iii. has documented one negative serum pregnancy test within 14 days prior to study entry.

5. The subject is willing to abstain from application of non-study topical medications to the skin of the face for the duration of the study, including prescription and over the counter preparations.

6. The subject is willing not to have targeted BCCs treated by their PSCP unless the BCCs are documented by Study Investigators, preferably on two separate visits, except when the PSCP believes that delay in treatment potentially might compromise the health of the subject.

List of Exclusion Criteria:

1. The subject has used topical or systemic therapies that might interfere with the evaluation of the study medication during the study.
2. The subject has a history of hypersensitivity to any of the ingredients in the study medication formulations.
3. The subject is unable to return for follow-up tests.
4. The subject has uncontrolled systemic disease, including known HIV positive patients.
5. The subject has a history of other skin conditions or significant illness that would interfere with evaluation of the study medication.
6. Any condition or situation which in the Investigator's opinion may put the subject at significant risk, could confound the study results, or could interfere significantly with the subject's participation in the study.
7. The subject has a history of invasive cancer within the past five years excluding non-melanoma skin cancer, Stage I cervical cancer, or CLL Stage 0.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-07; Primary Completion 2012-06 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ervin Epstein, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland; David R. Bickers, MD, Principal Investigator — Herbert Irving Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Children's Hospital Oakland Research Institute, Oakland, California
  - Children's Hospital Oakland Research Institiute, Oakland, California
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: 0.1% tazarotene cream first, then placebo
- Arm II: Vehicle (placebo) first, then 0.1% tazarotene cream
Period: First Intervention (12 Months)
Arm/Group | Arm I | Arm II
Started | 5 | 29
Completed | 2 | 25
Not Completed | 3 | 4
Period: Second Intervention (24 Months)
Arm/Group | Arm I | Arm II
Started | 2 | 25
Completed | 2 | 16
Not Completed | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients apply 0.1% tazarotene cream on months 0-12 and vehicle (placebo) on months 13-36 once daily to the chest.
  placebo : Applied to the skin
  tazarotene : Applied to the skin
- Arm II: Patients apply, vehicle (placebo) on months 0-12 and 0.1% tazarotene cream on months 13-36 once daily to the chest.
  placebo : Applied to the skin
  tazarotene : Applied to the skin
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 5 | 29 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 29 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (7) | 51 (13) | 53 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 14 | 17
  Male | 2 | 15 | 17
Region of Enrollment [Number; unit: participants]
  United States | 5 | 29 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction in the Observed Numbers of Basal Cell Carcinomas ≥ 9 mm² in Diameter
Time Frame: Baseline and 36 months
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 5 | 29
participants | 5 | 29

2. Primary Outcome: Parameters of Safety: Number of Participants With Adverse Events According to NCI CTCAE v3.0
Time Frame: Baseline and 36 months
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 5 | 29
participants | 5 | 29

ADVERSE EVENTS:
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 0/5 | 2/29
Other Adverse Events (participants affected / at risk) | 5/5 | 26/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=5) | Arm II (N=29)
prostate cancer diagnosis (Renal and urinary disorders) | 0 | 1
cellulitis and maxillary sinusitis (Ear and labyrinth disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=5) | Arm II (N=29)
Dryness (Skin and subcutaneous tissue disorders) | 0 | 6
Inflammation (Skin and subcutaneous tissue disorders) | 1 | 0
Itching (Skin and subcutaneous tissue disorders) | 0 | 3
Irritation (Skin and subcutaneous tissue disorders) | 2 | 4
Peeling (Skin and subcutaneous tissue disorders) | 0 | 4
Edema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4

LIMITATIONS AND CAVEATS:
Non-compliance and large drop-out rates leading to small numbers of data analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes